CLINICAL TRIAL: NCT06913309
Title: The Efficacy and Feasibility of Bright Light Therapy in Adolescents With Depressive Disorder: a Multi-center Randomized Controlled Double-blind Study
Brief Title: The Efficacy and Feasibility of Bright Light Therapy in Adolescents With Depressive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Collaborators: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiaozhen LV, Senior Researcher, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRWEP2024W074110106
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder，Major; Bright Light Therapy; Adolescent; Functional Neuroimaging; RCT
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bright light therapy（Light intensity is 10,000lux） (Experimental): In this study, participants randomly assigned to the intervention group will receive bright white light therapy interventions with light intensities of 10000 lux. The intervention plan is to receive 40 minutes of light therapy from 7:00-9:30 in the morning for 4 consecutive weeks, 6 days a week. The subject sits at a distance of 60cm from the light source.
  Interventions: Device: Bright light therapy（High light intensity）
- Bright light therapy（Light intensity is 5,000lux） (Experimental): In this study, participants randomly assigned to the intervention group will receive bright white light therapy interventions with light intensities of 5000 lux. The intervention plan is to receive 40 minutes of light therapy from 7:00-9:30 in the morning for 4 consecutive weeks, 6 days a week. The subject sits at a distance of 60cm from the light source.
  Interventions: Device: Bright light therapy（Low light intensity）
- Dim red light control intervention (Placebo Comparator): In this study, participants randomly assigned to the placebo-controlled group will receive dim red light therapy interventions with light intensities of 100 lux. The placebo-controlled intervention plan is to receive 40 minutes of red light therapy from 7:00-9:30 in the morning for 4 consecutive weeks, 6 days a week. The subject sits at a distance of 60cm from the light source.
  Interventions: Device: Dim red light placebo-controlled intervention

INTERVENTIONS:
Device: Bright light therapy（High light intensity） — In this study, we will utilize the optocoupler-controllable light source, a product jointly developed by the School of Physics at Peking University and Peking University Sixth Hospital, which granted a national patent in China, for the purpose of intervention.
  Participants randomly assigned to the high light density intervention group will receive bright white light therapy interventions with light intensities of 10000 lux, and the main wavelength of light source is 476.4nm. The intervention plan is to receive 40 minutes of light therapy from 7:00-9:30 in the morning for 4 consecutive weeks, 6 days a week. The subject sits at a distance of 60cm from the light source.
  Arms: Bright light therapy（Light intensity is 10,000lux）
Device: Bright light therapy（Low light intensity） — In this study, we will utilize the optocoupler-controllable light source, a product jointly developed by the School of Physics at Peking University and Peking University Sixth Hospital, which granted a national patent in China, for the purpose of intervention. Participants randomly assigned to the low light density intervention group will receive bright white light therapy interventions with light intensities of 5,000 lux,and the main wavelength of light source is 476.4nm. The intervention plan is to receive 40 minutes of light therapy from 7:00-9:30 in the morning for 4 consecutive weeks, 6 days a week. The subject sits at a distance of 60cm from the light source.
  Arms: Bright light therapy（Light intensity is 5,000lux）
Device: Dim red light placebo-controlled intervention — In this study, participants randomly assigned to the placebo-controlled group will receive dim red light therapy interventions with light intensities of 100 lux, and the main wavelength of light source is 690.4nm. The placebo-controlled intervention plan is to receive 40 minutes of red light therapy from 7:00-9:30 in the morning for 4 consecutive weeks, 6 days a week. The subject sits at a distance of 60cm from the light source.
  Arms: Dim red light control intervention

SUMMARY:
Major Depressive Disorder (MDD) is a chronic disease characterized by a high prevalence, low cure rate, and significant disability. Globally, depression is recognized as the leading cause of illness and disability among children and adolescents aged 10 to 19 years. Bright light therapy has been established as an effective treatment for seasonal affective disorder and has demonstrated considerable efficacy in adult patients with major depressive disorder. However, its application in adolescent patients with major depressive disorder remains largely unexplored. The aim of this clinical trial is to evaluate the efficacy and feasibility of bright light therapy in adolescents with major depressive disorder and to explore the potential neural mechanisms by which bright light therapy enhances emotional and cognitive function in this population. This is a multicenter, randomized, controlled, double-blind study. It will involve adolescents aged 13 to 17 who are either untreated or have been stable on medication for at least one week. Adolescents with major depressive disorder will be randomly assigned to one of three groups: a high-intensity bright light intervention group, a low-intensity bright light intervention group, and a control group receiving dark red light. Each group will undergo four weeks of light exposure, six days per week, for 40 minutes daily between 7:00 and 9:30 AM. During the light exposure period, follow-up assessments will be conducted every weekend, and participants will be followed for two weeks after the completion of light exposure.

Additionally, the study will include healthy adolescent controls and collect functional Near-Infrared Spectroscopy (fNIRS) data from both the adolescent participants with major depressive disorder and the healthy controls at baseline. The fNIRS data will also be collected from the adolescent participants with major depressive disorder at the end of the intervention, in order to investigate the potential neural mechanisms by which light therapy alleviates depressive symptoms in adolescents.

ELIGIBILITY:
1. Adolescents with Major Depressive Disorder

   Inclusion Criteria:all of the following conditions were met for inclusion:
   * Meet the diagnostic criteria for depressive episodes in the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) (either first or recurrent), and be clearly diagnosed by two physicians using MINI-kid 2.0;

     * Age 13 to 17 years, right-handed, and gender-neutral; ③Not currently on medication; or have been stabilized on the original medication regimen for at least 1 week; ④ Hamilton Depression Scale (HAMD-17) score ≥14 at baseline; ⑤ Years of education ≥ 5 years and can cooperate in completing the scale assessment;

       * Subjects volunteered to participate in the study, and both subjects and guardians signed an informed consent form.

   Exclusion Criteria: excluded if any of the following conditions are met:
   * A history of previous or current episodes of other psychiatric disorders, such as (schizophrenia, autism spectrum disorders, and schizoaffective disorders, etc.);

     * Previous history of drug or substance abuse or dependence;

       * Total score of ≥ 8 on the Young's Mania Scale as assessed by the investigator for the subject;

         ④ Have received, or are currently receiving, or have planned to receive in the last month, other systemic interventions other than medication in the 6 months prior to enrollment, e.g., systemic psychotherapy (1 to 2 times per month for more than 6 months), physical therapy other than phototherapy, or exercise therapy;

         ⑤ Those who are medically unstable, or unable to cooperate in completing the study; those who are currently at serious risk of suicide as assessed by the investigator (HAMD-17 entry 3 score ≥ 3);
         * Comorbid serious physical illnesses such as severe liver function abnormalities, hyper/hypothyroidism and abnormal thyroid function, encephalitis, head trauma or coma, epilepsy, loss of consciousness, diabetes mellitus, renal failure, etc.; or those whose clinical laboratory findings at the time of enrollment are, in the opinion of the investigator, significantly out of the reference range and of clinical significance; ⑦ Comorbid visual pathway diseases (retinal detachment, optic nerve atrophy, macular degeneration, etc.), systemic diseases that have an impact on the retina, high myopia (myopia of 600 degrees and above); or those who are using photosensitizers, drugs with potential photosensitizing effects (e.g., chlorpromazine, tricyclic antidepressant, chrysothema, etc.); ⑧ According to the opinion of the research group, those who are not suitable for other conditions of this study.
2. Adolescent Health Controls

   Criteria for inclusion: All of the following conditions were met for inclusion:
   * Age 13-17 years old, right-handed, gender is not limited;

     * Years of education ≥ 5 years, can cooperate with the completion of the scale assessment; ③Subjects volunteered to participate in the study, and both subjects and guardians signed an informed consent form.

   Exclusion Criteria: excluded if any of the following conditions are met:

   ①Previous or current suffering from any mental illness (e.g., schizophrenia, loneliness spectrum disorders, anxiety disorders and schizoaffective disorders, etc.), or a history of drug or substance abuse or dependence;

   ② First-degree relatives with a family history of mental illness;

   ③Comorbid serious physical illnesses such as severe liver function abnormalities, hyper/hypothyroidism and thyroid function abnormalities, encephalitis, head trauma or coma, epilepsy, loss of consciousness, diabetes mellitus, renal failure, etc.; or those whose clinical laboratory findings at the time of enrollment were considered by the investigator to be significantly out of the reference range and of clinical significance;

   ④ Those with other conditions that, according to the opinion of the study group, are not suitable for this study.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale-17 | baseline，7 days after the intervention begin，14 days after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  The Hamilton Depression Rating Scale-17 (HAMD-17), developed by Hamilton in 1960, is a widely used clinical rating scale consisting of 17 items that evaluate various depressive symptoms, including mood, suicidal thoughts, sleep disturbances, loss of interest, psychomotor changes, anxiety, gastrointestinal and somatic symptoms, sexual dysfunction, and weight loss. Scored on a scale of 0 to 4 (with some items possibly using a 0 to 2 scale), the total score reflects the severity of depressive symptoms and is used for diagnosing depression, planning tailored treatment, monitoring treatment effectiveness, and conducting research on depression treatment efficacy.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 | baseline，7 days after the intervention begin，14 days after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  The Generalized Anxiety Disorder-7 is a standardized assessment tool developed by Spitzer et al. in 2006. It is a 7-item questionnaire designed to evaluate the severity of anxiety symptoms over the past two weeks. The scale covers various aspects of anxiety, including feelings of tension, worry, irritability, and difficulty relaxing. Each item is rated on a 4-point scale, ranging from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21. Higher scores indicate more severe anxiety symptoms. The GAD-7 is primarily used as a screening and assessment tool in clinical and research settings, aiding clinicians in identifying and quantifying anxiety symptoms, monitoring changes over time, and evaluating treatment effectiveness. It is a simple, reliable, and valid instrument that can be easily administered and scored, making it a valuable addition to the clinical assessment of anxiety disorders.
Quick Inventory of Depressive Symptomatology-Self-Report | baseline， every day of the first two weeks after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  The Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR16), a rigorous and systematic self-assessment scale developed by Rush et al. in 2003 with subsequent refinements, is a widely recognized tool for quickly gauging depressive symptoms over the past week. It comprises 16 items covering various dimensions of depression, including mood, sleep, appetite, energy levels, concentration, self-esteem, suicidal ideation, and daily functioning, each rated on a 4-point scale (0-3). The scale assesses the severity and frequency of symptoms, with higher scores indicating more severe depression. The QIDS-SR16 serves multiple purposes: it aids in screening and assessing depressive symptoms in clinical settings, allows individuals to monitor their depressive state over time, serves as a research tool in clinical studies evaluating treatment effectiveness, and provides valuable information that can support the diagnostic process when combined with clinical interviews.
Pittsburgh Sleep Quality Inventory | baseline，7 days after the intervention begin，14 days after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  The PSQI, or Pittsburgh Sleep Quality Inventory, was developed by Buysse et al. in 1989. It is a widely used and standardized self-report questionnaire designed to assess sleep quality over the past month. The PSQI consists of 19 self-rated items and 5 additional items for bed partner or roommate ratings (though only 18 of the self-rated items are scored). The assessment covers seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored on a 0-to-3 scale, with the total PSQI score ranging from 0 to 21. Higher scores indicate poorer sleep quality, with a total score of 5 or less indicating good sleep quality, 6-10 indicating fair sleep quality, 11-15 indicating poor sleep quality, and 16 or more indicating very poor sleep quality. The PSQI serves multiple purposes, including clinical diagnosis of sleep disorders, research on sleep quality, and eval
Hopkins Verbal Learning Test-Revised | baseline, 7 days after the intervention begin，14 days after the intervention begin, 28 days after the intervention begin，14 days after the intervention accomplished
  Hopkins Verbal Learning Test-Revised (HVLT-R) is a widely used neuropsychological assessment tool designed to evaluate verbal memory and cognitive function. Developed by J. Brandt and Benedict in 2001, the HVLT-R consists of a list of 12 nouns divided into three semantic categories (e.g., dwelling places, four-legged animals, and precious stones), with four words per category. The assessment involves three learning trials, where participants are presented with the list of words and are asked to recall as many words as possible immediately after each presentation. Additionally, there is a delayed recall trial, where participants are asked to recall the words after a delay of 20-25 minutes. The scoring principle is based on the number of correctly recalled words during each learning trial and the delayed recall trial. The total score for the three learning trials and the delayed recall trial is calculated, as wel
Brief Visuospatial Memory Test-Revised | baseline，7 days after the intervention begin，14 days after the intervention begin，28 days after the intervention begin，14 days after the intervention accomplished
  Brief Visuospatial Memory Test-Revised is a neuropsychological assessment tool designed to evaluate visual spatial memory. Developed by researchers including Barr, Morrison, Zaroff, and Devinsky in 2004, the BVMT-R consists of six geometric figures presented in a 2x3 array, serving as the stimuli for the test. The assessment involves three learning trials, where participants are shown the stimuli for 10 seconds and are then asked to draw as many of the figures as possible in the correct locations on a response sheet. After a delay of approximately 25 minutes, a delayed recall trial is administered, followed by a recognition trial where participants are asked to identify the original geometric figures among a set of 12. The scoring principle is based on the number of correctly recalled and recognized figures. It provides valuable information for diagnosing, monitoring disease progression, and evaluating the effectiveness of interventions.
Trail Making Test | baseline，7 days after the intervention begin，14 days after the intervention begin，28 days after the intervention begin，14 days after the intervention accomplished
  The Trail Making Test (TMT）is divided into two parts, A and B. Each part consists of a practice and a test. The TMT-A requires the examinee to complete the lines from 1 to 25 in smallest-to-largest order as fast as possible, without taking the pen off the paper, while the TMT-B requires the examinee to complete the lines from 1 to 25 in smallest-to-largest order, with circle icons and square icons spaced out as fast as possible, without taking the pen off the paper. The pen is not allowed to leave the paper surface during the process of connecting the lines. Record the time taken for each of the two parts. Cut-off values: TMT-A: 50-59 years old: less than 70 seconds; 60-69 years old: less than 80 seconds; 70-79 years old: less than 100 seconds; TMT-B: 50-59 years old: 180 seconds; 60-69 years old: 200 seconds; 70-79 years old: 240 seconds. The shorter the time, the better the executive function.
  Translated with DeepL.com (free version)
The General Self-Efficacy Scale | baseline，7 days after the intervention begin，14 days after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  The General Self-Efficacy Scale (GSES) is a psychological assessment tool with its roots in the self-efficacy theory developed by Ralf Schwarzer. First compiled by Schwarzer and his colleagues at Freie Universität Berlin in 1981 (with later refinements leading to a 10-item version), the GSES measures an individual's confidence and belief in their ability to successfully complete tasks or cope with challenges across various situations. It consists of 10 items that assess facets of self-efficacy, such as confidence in facing complex tasks, problem-solving abilities, persistence in overcoming difficulties, and a sense of control over future outcomes. The scale employs a Likert-type 4-point rating system, where respondents indicate their agreement with each statement on a scale from 'completely incorrect' (scored as 1) to 'completely correct' (scored as 4).The total score provides a measure of general self-efficacy, with higher scores indicating stronger self-efficacy.
Young Mania Rating Scale | baseline，7 days after the intervention begin，14 days after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  The Young Mania Rating Scale (YMRS), developed by R.C. Young and colleagues in 1978, is a clinician-administered rating scale designed to assess the severity of manic symptoms over the past week. It comprises 11 items that evaluate various aspects of mania, including elevated mood, increased activity and energy, sexual interest, sleep pattern, irritability, speech, language-thought disorders, content of thought, aggressive or destructive behavior, appearance, and insight. The scoring system varies across items, with some rated on a 0-4 scale and others on a 0-8 scale. The total score is obtained by summing the ratings of all items, providing a quantitative measure of manic severity. Higher scores indicate more severe manic symptoms. The YMRS is primarily used in clinical and research settings for the assessment of manic states.
Asberg Side-Effect Rating Scale for Antidepressants | baseline，7 days after the intervention begin，14 days after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  Asberg Side-Effect Rating Scale for Antidepressants (SERS) is a rating scale developed by Swedish psychiatrist M. Asberg in 1970. It is specifically designed to evaluate the adverse effects experienced by individuals following the administration of antidepressant medications. The scale contains 14 items that assess a wide range of symptoms, including physical fatigue, dizziness, headache, sleep disturbance, orthostatic hypotension, palpitations, tremors, sweating, dry mouth, constipation, urinary difficulties, somnolence, sexual dysfunction, and other symptoms. Each item is rated on a 4-point scale ranging from 0 (absent) to 3 (severe), allowing for a comprehensive quantification of the severity of side effects. The total score, calculated by summing the ratings of all items, provides an overall measure of antidepressant-related adverse effects. The SERS is primarily used in clinical and research settings to aid in the identification, monitoring, and documentation of side effects.
Adolescent Irritability Rating Scale | baseline，7 days after the intervention begin，14 days after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  The Adolescent Irritability Rating Scale (ARI) is a standardized assessment tool designed to measure the degree of irritability in adolescents. The ARI scale was created as a measure of parent and self-assessment.It was developed by experts in the field of psychology and psychiatry, though specific authorship and the year of its development may vary depending on the version or update. The scale typically includes multiple items that comprehensively evaluate various aspects of irritability, such as the frequency and intensity of anger outbursts, reactions to minor frustrations, and the duration and consistency of irritable mood. Each item is scored on a specific rating scale, often ranging from 0 (indicating no irritability) to a higher number (reflecting increasing levels of irritability), allowing for a quantitative analysis of irritability severity. The total score, obtained by summing the ratings of all items, provides an overall measure of irritability in adolescents.
Morningness-Eveningness Questionnaire-Self-Assessment | baseline，14 days after the intervention begin，28 days after the intervention begin，14 days after the intervention accomplished
  The Morningness-Eveningness Questionnaire-Self-Assessment (MEQ-SA) is a widely-used self-rating tool designed to measure individual differences in circadian rhythm types, specifically distinguishing between "morning types" (also known as "larks") and "evening types" (also known as "owls").Each item on the MEQ-SA is scored on a specific scale, with the total score being the sum of all individual item scores. The scoring range typically varies from 16 to 86, with lower scores indicating a stronger tendency towards eveningness and higher scores suggesting a morningness predisposition. Specifically, scores of 41 or below are classified as "evening type," scores between 42 and 58 are considered "intermediate," and scores of 59 or above are categorized as "morning type."
The Seasonal Pattern Assessment Questionnaire | baseline
  The Seasonal Pattern Assessment Questionnaire (SPAQ) is a comprehensive evaluation tool designed to assess the seasonal variations in various aspects of an individual's life, including sleep, social interactions, mood, weight, appetite, and energy levels.Each item on the SPAQ is scored on a specific scale, reflecting the degree to which the individual experiences seasonal variations in the respective domain. The total score, derived from the summation of individual item scores, provides an overall measure of seasonal pattern intensity. The scoring principles are designed to ensure that higher scores indicate more pronounced seasonal variations.
Stroop Color-Word Test | baseline，7 days after the intervention begin，14 days after the intervention begin， 28 days after the intervention begin， 14 days after the intervention accomplished
  The Stroop Color Word Test (CWT) was developed by Professor Stroop in 1935 to evaluate subjects' executive functions. The test is a measure of selective attention and the degree of inhibition of irrelevant information in executive functioning. It consists of three main parts: reading words (Stroop-w), color naming (Stroop-c), and color-word interference (Stroop-cw), which require subjects to accurately and quickly read the words or the colors, respectively, as required.
Ottawa Self-Injury Inventory | baseline，7 days after the intervention begin，14 days after the intervention begin，21 days after the intervention begin，28 days after the intervention begin，7 days after the intervention accomplished，14 days after the intervention accomplished
  The Ottawa Self-Injury Inventory (OSI), a revision of the Quinn Self-Injury Questionnaire (1998) by Cloutier et al. is a more comprehensive assessment tool for assessing NSSI behaviors. It includes the frequency of actual NSSI behaviors, suicide attempts, visits to the doctor after self-injury, the source of the first self-injurious thoughts, the mode and location of self-injury, and methods of resisting self-injury. The Functional Scale section included the Self-Injury Motivation and Addiction Characteristics scales.Martin's factor analysis of the Motivation section of the scale revealed that it consisted of 4 factors, Internal Emotion Regulation, Social Influence, External Emotion Regulation, and Stimulus Seeking, each of which was scored on a 5-point scale from 0 (never) to 4 (always), with the higher the score, the higher the level of motivation. The Addiction Characteristics section consists of 7 individual items, each of which is scored on a 5-point scale from 0 (never) to 4 (al

IPD SHARING:
Plan to Share IPD: Undecided